CLINICAL TRIAL: NCT00924677
Title: Phase 1 Study of Therapeutic Methods for Chronic Knee Osteoarthritis Pain
Brief Title: The Effect of Therapeutic Methods for Chronic Knee Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Jinwoo Shin, anesthesiology and pain medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN0901
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Osteoarthritis, Knee
Keywords: genicular nerve; osteoarthritis; knee; neurotomy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocaine (Sham Comparator): Local injection with lidocaine through the RF cannula without activation of RF generator.
  Interventions: Procedure: radiofrequency neurotomy sham therapy
- lidocaine, radiofrequency current (Active Comparator): After lidocaine injection through the RF cannula, the temperature of the electrode tip was raised to 70℃ for 90 seconds by RF generator.
  Interventions: Procedure: radiofrequency neurotomy for genicular nerve

INTERVENTIONS:
Procedure: radiofrequency neurotomy for genicular nerve — RF cannula was advanced percutaneously towards areas connecting the shaft to epicondyle of femur or tibia. Lidocaine (1 mL of 2%) was injected before activation of the RF generator (NeuroThermTM, Morgan automation LTD, Liss, UK). RF electrode was inserted through RF cannula. The temperature of the electrode tip was raised to 70℃ for 90 seconds by radiofrequency generator.
  Other Names: neuroablation or radiofrequency neurolysis
  Arms: lidocaine, radiofrequency current
Procedure: radiofrequency neurotomy sham therapy — The placebo (sham) group received the same procedure without activation of the RF generator.
  Other Names: radiofrequency neurolysis sham therapy
  Arms: lidocaine

SUMMARY:
Chronic osteoarthritis (OA) pain of the knee is not effectively abrogated by the available non-pharmacologic or pharmacologic treatments. Radiofrequency (RF) neurotomy is a therapeutic alternative for chronic pain. Here, the researchers investigate the efficacy of RF neurotomy applied to articular branches (genicular nerves) in treating knee joint pain.

DETAILED DESCRIPTION:
The knee joint is innervated by articular branches of various nerves (femoral, common peroneal, saphenous, tibial and obturator) (Kennedy et al. 1982; Hirasawa et al. 2000). These articular branches around the knee joint are known as genicular nerves. Several genicular nerves can be easily approached percutaneously under fluoroscopic guidance. In our study, genicular nerves were effectively blocked with local anesthetics under fluoroscopic guidance, leading to a significant reduction in knee pain. Rf neurotomy is based on the theory that cutting the nerve supply to a painful structure may alleviate pain and restore function. we evaluate the efficacy of RF neurotomy in reducing pain and improving function in the elderly with chronic knee OA.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic knee pain (i.e., knee pain of moderate intensity or greater on most or all days for ≥ 3 months)
* patients with radiologic knee osteoarthritis (Kellgren-Lawrence grade 2-4, evaluated by a radiologist)

Exclusion Criteria:

* acute knee pain
* prior knee surgery
* other connective tissue diseases affecting the knee
* serious neurologic or psychiatric disorders
* injection with steroids or hyaluronic acids during the previous 3 months
* sciatic pain
* anticoagulant medications
* pacemakers
* prior electroacupuncture treatments

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale pain scores | at 12 weeks after the procedure

SECONDARY OUTCOMES:
Oxford knee score | at 12 weeks after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pyong-hwan Park, M.D., Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Kennedy JC, Alexander IJ, Hayes KC. Nerve supply of the human knee and its functional importance. Am J Sports Med. 1982 Nov-Dec;10(6):329-35. doi: 10.1177/036354658201000601. PMID 6897495
- [Result] van Kleef M, Barendse GA, Kessels A, Voets HM, Weber WE, de Lange S. Randomized trial of radiofrequency lumbar facet denervation for chronic low back pain. Spine (Phila Pa 1976). 1999 Sep 15;24(18):1937-42. doi: 10.1097/00007632-199909150-00013. PMID 10515020